CLINICAL TRIAL: NCT06621316
Title: To Explore the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Multiple Doses of HRS-7535 in Obese Subjects
Brief Title: A Study of Safety and Tolerability of Multiple Doses of HRS-7535 in Obese Subjects
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7535-107
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo parallel-controlled Ib/II clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Treatment group A (Experimental): HRS-7535 Tablet at dose level 1
  Interventions: Drug: HRS-7535 Tablet
- Treatment group B (Experimental): HRS-7535 Tablet at dose level 2
  Interventions: Drug: HRS-7535 Tablet
- Treatment group C (Experimental): HRS-7535 Tablet at dose level 3
  Interventions: Drug: HRS-7535 Tablet
- Treatment group D (Experimental): HRS-7535 Tablet at dose level 4
  Interventions: Drug: HRS-7535 Tablet
- Treatment group E (Placebo Comparator): Placebo at dose level 1
  Interventions: Drug: Placebo
- Treatment group F (Placebo Comparator): Placebo at dose level 2
  Interventions: Drug: Placebo
- Treatment group G (Placebo Comparator): Placebo at dose level 3
  Interventions: Drug: Placebo
- Treatment group H (Placebo Comparator): Placebo at dose level 4
  Interventions: Drug: Placebo
- Treatment group I (Experimental): HRS-7535 Tablet at dose level 1 or level 2 or level 3 or level 4.
  Interventions: Drug: HRS-7535 Tablet
- Treatment group J (Experimental): HRS-7535 Tablet at dose level 1 or level 2 or level 3 or level 4.
  Interventions: Drug: HRS-7535 Tablet
- Treatment group K (Placebo Comparator): Placebo at dose level 1 or level 2.
  Interventions: Drug: Placebo
- Treatment group L (Placebo Comparator): Placebo at dose level 1 or level 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-7535 Tablet — at multiple dose levels
  Arms: Treatment group A; Treatment group B; Treatment group C; Treatment group D; Treatment group I; Treatment group J
Drug: Placebo — at multiple dose levels (matching active arm HRS-7535 Tablet)
  Arms: Treatment group E; Treatment group F; Treatment group G; Treatment group H; Treatment group K; Treatment group L

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple doses of HRS-7535 tablet in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. At screening: BMI ≥30 kg/m2.
3. Have been controlled by diet and exercise for 3 months or more before screening, and the change in body weight in the past 3 months is less than 5%.
4. Male and female subjects of childbearing potential through signing the informed consent form to 1 month after the last dose have no family plans and must use highly effective contraception, and female participants of childbearing potential also must have no plans to donate eggs (male participants must have no plans to be sperm donors); Female subjects of childbearing potential must have a serum pregnancy test within 7 days prior to the date of randomization, including the day of randomization.

Exclusion Criteria:

1. Clinically significant abnormalities in relevant laboratory tests at screening.
2. The results of the electrocardiogram at screening show clinically significant abnormalities that may affect the safety of the subject, including but not limited to myocardial infarction, severe arrhythmias such as supraventricular tachycardia, atrial fibrillation, atrial flutter, second- or third-degree atrioventricular block, etc.
3. Heart rate or pulse > 100 beats per minute or ECG QTcF >450 ms at screening.
4. The PHQ-9 score ≥ 15 points.
5. Poor blood pressure control at screening.
6. Presence or history of endocrine disease that may significantly affect body weight at screening.
7. History of diabetes mellitus.
8. Within 6 months prior to screening, the subject has the following diseases of clinical significance: including but not limited to neurological, psychiatric, cardiovascular, endocrine, gastrointestinal, respiratory, urinary, blood, immune system and other diseases, which may interfere with the trial results or pose additional risks to the administration of the study drug as judged by the investigator.
9. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
10. Previous or known history of acute or chronic pancreatitis, history of cholecystitis or history of gallstones, chronic malabsorption syndrome or cholestasis.
11. Severe cardiovascular and cerebrovascular diseases within 6 months prior to screening, including but not limited to: heart failure (NYHA grade II-IV), angina, stroke or transient ischemic attack, myocardial infarction, severe arrhythmia, or coronary artery bypass grafting or percutaneous coronary intervention, etc.; and/or planned revascularization of the coronary arteries, carotid arteries, or peripheral arteries at the time of screening.
12. Any malignant tumor of any organ system within 5 years, regardless of whether there is evidence of local recurrence or metastasis, except for cured local cancer, such as: local basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the prostate.
13. Those who have had serious infections, severe trauma, major and medium-sized surgeries, or planned to undergo surgery during the trial within 6 months prior to screening.
14. Those with or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia or other more serious mental illness; or mentally incapacitated or with a language impairment that is unable to fully understand the trial protocol or is unwilling to collaborate with study center staff.
15. Presence of a history of acute or chronic hepatitis or other serious liver disease other than non-alcoholic fatty liver disease.
16. Presence of any blood disorder (e.g., hemolytic anemia, sickle cell disease, etc.) that may interfere with HbA1c detection.
17. Autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis).
18. Use of medications or treatments that may cause significant weight gain or loss within 2 months prior to screening:

    * glucocorticoids (short-term systemic use< 7 days or topical, inhaled, intraocular and nasal administration);
    * tricyclic antidepressants, atypical antipsychotics and mood stabilizers (such as imipramine, chlorpromazine, amitriptyline, mirtazapine, clozapine, olanzapine, paroxetine, phenelzine, thioridazine, valproic acid and its derivatives, lithium salts, etc.);
    * Orlistat, GLP-1 receptor agonists, or incretins, or other weight-loss therapies other than diet and exercise (including GLP-1 receptor agonists, multi-targeted agents);
    * Other medications or treatments that may significantly affect blood sugar or body weight (eg, metformin, SGLT-2 inhibitors, etc.).
19. Undergoing or planning bariatric surgery or weight-loss therapy based on endoscopy and/or medical devices, etc. during the study period (except for a history of liposuction surgery greater than 1 year).
20. Prior discontinuation of GLP-1 receptor agonist-containing agents for safety and/or tolerability reasons.
21. whichever is longer: Participated in a clinical trial of any drug or medical device within 3 months prior to screening or is still within 5 half-lives of the investigational drug. Participation in clinical trials is defined as: signing informed consent and using investigational drugs (including placebo) or investigational medical devices; Participated in clinical trials of drugs containing GLP-1 receptor agonists (including placebo) within 6 months prior to screening.
22. Known or suspected hypersensitivity to GLP-1 receptor agonist drugs, the investigational drug or its components, or its excipients.
23. Addiction to tobacco and alcohol.
24. Those who have a history of blood donation or blood loss of ≥400ml within 3 months before screening or have received blood transfusion within 2 months.
25. Subjects who are mentally incapacitated or have language impairment who cannot fully understand or participate in the trial process.
26. Females who are pregnant, lactating, planning to become pregnant during the trial, or subjects of childbearing potential who are unwilling to use highly effective contraception during the trial period (starting from signing the informed consent form) and within 1 month after the last dose.
27. Inability to tolerate venipuncture blood sampling or needle phobia.
28. Any condition judged by the investigator to be unsuitable to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 24 weeks

SECONDARY OUTCOMES:
Pharmacokinetic endpoint: Concentration of HRS-7535 in plasma | 24 weeks
Change in fasting weight at week 24 | 24 weeks
Change in waist circumference at week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Peoples Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided